CLINICAL TRIAL: NCT07218315
Title: Nanosecond Pulsed Field Ablation in the Management of T1N0M0 Papillary Thyroid Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0726; NCI-2025-07697 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with nsPFA (Experimental): Participants will undergo thyroid ablation with the CellFX nsPFA system, an outpatient procedure under local anesthesia, or intravenous sedation.
  Interventions: Device: CellFX nsPFA Percutaneous Electrode System

INTERVENTIONS:
Device: CellFX nsPFA Percutaneous Electrode System — Patients will undergo thyroid ablation with the CellFX nsPFA system, an outpatient procedure under local anesthesia, or intravenous sedation.

SUMMARY:
This study is to evaluate the effectiveness of nsPFA in treating papillary thyroid microcarcinoma. T

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the efficacy of ultrasound-guided nsPFA™ in the treatment of patients with T1N0M0 PTC as measured by the thyroid nodule volume changes including volume reduction rate (VRR), technique efficacy (TE) and nodule regrowth (NR) during post procedure follow-up.

Secondary Objectives:

To assess the clinical safety and complications of the CellFX Percutaneous Electrode (PE) System

To evaluate the ultrasound features of thyroid nodules over time following ultrasound-guided nsPFA.

To determine the health-related quality of life changes over time induced by ultrasound-guided nsPFA.

ELIGIBILITY:
Inclusion Criteria:

* Participant must provide voluntary, written informed consent to participate in this clinical investigation.
* Participant agrees to comply with all study procedures, including all follow-up visits.
* Participant with a Bethesda VI cytology (tumor size <= 1.5 cm, no known regional/distant metastases)
* Participant with a Bethesda V cytology and normal calcitonin levels.
* Ultrasonographic evaluation of tumor to be ablated must show size of less than or equal to 1.5 cm and no extrathyroidal extension or locoregional metastases.
* Participant must have normal complete blood count, blood coagulation profile, and thyroid function test.
* For females of childbearing potential, a negative serum or urine pregnancy test must be obtained at baseline, prior to the procedure.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following: ). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
  * History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study procedure.

Exclusion Criteria:

* FNA findings suggestive of high-grade malignancy
* Presence of regional or distant lymph node metastases.
* Participant had a history of previous neck irradiation.
* Females who are pregnant at time of enrollment.
* Participant has any condition or situation, in the opinion of the site Investigator, that puts the subject at significant risk, could confound the study results, or may interfere significantly with subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Victoria E Banuchi, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org